CLINICAL TRIAL: NCT02426021
Title: A Phase 1, Single-Dose Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Subcutaneous Injection of MLN1202 in the Japanese and Caucasian Healthy Male Participants
Brief Title: Phase 1 Single Subcutaneous Dose Study of MLN1202
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision; No Safety or Efficacy Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN1202/CPH-001; U1111-1169-0038 (Registry Identifier: UTN); JapicCTI-152874 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-04-21; First posted 2015-04-24 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Healthy Japanese and Caucasian Male Adults
MeSH Terms: interventions — plozalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort J1: MLN1202 (75 mg) (Experimental): Single subcutaneous administration of MLN1202 (75 mg) in 6 healthy Japanese male adults
  Interventions: Drug: MLN1202
- Cohort J1: placebo (Experimental): Single subcutaneous administration of placebo in 2 healthy Japanese male adults
  Interventions: Drug: MLN1202 Placebo
- Cohort J2:MLN1202 (105 mg) (Experimental): Single subcutaneous administration of MLN1202 (105 mg) in 6 healthy Japanese male adults
  Interventions: Drug: MLN1202
- Cohort J2: placebo (Experimental): Single subcutaneous administration of placebo in 2 healthy Japanese male adults
  Interventions: Drug: MLN1202 Placebo
- Cohort J3: MLN1202 (150 mg) (Experimental): Single subcutaneous administration of MLN1202 (150 mg) in 6 healthy Japanese male adults
  Interventions: Drug: MLN1202
- Cohort J3: placebo (Experimental): Single subcutaneous administration of placebo in 2 healthy Japanese male adults
  Interventions: Drug: MLN1202 Placebo
- Cohort J4: MLN1202 (450 mg) (Experimental): Single subcutaneous administration of MLN1202 (450 mg) in 6 healthy Japanese male adults
  Interventions: Drug: MLN1202
- Cohort J4: placebo (Experimental): Single subcutaneous administration of placebo in 2 healthy Japanese male adults
  Interventions: Drug: MLN1202 Placebo
- Cohort C1: MLN1202 (75 mg) (Experimental): Single subcutaneous administration of MLN1202 (75 mg) in healthy Causacian male adults
  Interventions: Drug: MLN1202
- Cohort C2: MLN1202 (150 mg) (Experimental): Single subcutaneous administration of MLN1202 (150 mg) in healthy Causacian male adults
  Interventions: Drug: MLN1202

INTERVENTIONS:
Drug: MLN1202 — Subcutaneous administration of MLN1202
  Arms: Cohort C1: MLN1202 (75 mg); Cohort C2: MLN1202 (150 mg); Cohort J1: MLN1202 (75 mg); Cohort J2:MLN1202 (105 mg); Cohort J3: MLN1202 (150 mg); Cohort J4: MLN1202 (450 mg)
Drug: MLN1202 Placebo — Subcutaneous administration of MLN1202 placebo
  Arms: Cohort J1: placebo; Cohort J2: placebo; Cohort J3: placebo; Cohort J4: placebo

SUMMARY:
The objective of the study is to investigate the safety, pharmacokinetics, and pharmacodynamic effect of a single dose of MLN1202 in healthy Japanese male adults.

DETAILED DESCRIPTION:
This is a single dose, phase 1 study in healthy Japanese and Caucasian male adults.

Japanese subjects will be assigned to Cohort J1 (at a dose of 75 mg), Cohort J2 (105 mg), Cohort J3 (150 mg), or Cohort J4 (450 mg) in a randomized, double-blind, placebo-controlled manner, while Caucasian subjects to Cohort C1 (at a dose of 75 mg) or Cohort C2 (150 mg) in an open-label manner.

Takeda has made a business decision to terminate this study due to portfolio re-prioritization. There were no safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written informed consent form (ICF) prior to the initiation of any study procedures.
3. The participant is a healthy adult man who is defined as Japanese (all parents and grandparents of the participant are Japanese) or Caucasian (all parents and grandparents of the participant are Caucasian).
4. The participant is between 20 and 45 years of age at the time of informed consent.
5. The participant has a body weight of at least 50 kg and has a body mass index (BMI) between 18.5 and 25.0 kg /m2 when the participant is Japanese or between 18.5 and 30.0 kg /m2 when the participant is Caucasian at the time of screening and baseline examination.
6. A male participant who is sexually active with a female partner of childbearing potential and who has not received contraceptive therapy agrees to use adequate contraception from the time of informed consent until 12 weeks (84 days) after administration of the study drug.

Exclusion Criteria:

1. The participant has received any other investigational compound within 16 weeks (112 days) prior to administration of the study drug.
2. The participant has previously received agents containing MLN1202, a monoclonal antibody or monoclonal antibody fragment.
3. The participant has been vaccinated within 4 weeks (28 days) prior to administration of the study drug or is planning to be vaccinated during the study period.
4. The participant is a study site employee or immediate family member of the employee, or may consent under duress.
5. The participant has poorly-controlled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, or endocrine disease, hemorrhagic disorder or other abnormalities which may impact the ability of the participant to participate or potentially confound the study results.
6. The participant has recurrent serious or poorly-controlled infection and is considered to have difficulty participating in the study by the investigator.
7. The participant has a history of hypersensitivity or allergies to MLN1202 or additives contained in MLN1202 preparations.
8. The participant has a history of hypersensitivity or allergies to monoclonal antibodies other than MLN1202.
9. The participant has positive results in urine drug tests at screening.
10. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol dependence within 2 years prior to the study visit at screening or is unwilling to agree to abstain from alcohol and drugs throughout the study period.
11. The participant requires any excluded medication or food products listed in the Excluded Medications and Dietary Products (see section 7.3) during the study period.
12. The participant intends to donate sperm during the study period or period until 12 weeks (84 days) after administration of the study drug.
13. The participant has a history of cancer.
14. The participant has, is suspected of having, or has a history of active tuberculosis or latent tuberculosis infection.
15. The participant has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis B virus antibody (hepatitis B surface antibody [HBsAb]/ hepatitis B core antibody [HBcAb]), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at screening. This does not include the participant who has a positive test result only for HBsAb due to HBV vaccination.
16. The participant has used nicotine-containing products (cigarettes, pipes, cigars, chewing tobacco, nicotine patches, or nicotine gum, etc.) within 4 weeks (28 days) prior to administration of the study drug.
17. The participant has poor peripheral venous access.
18. The participant has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to administration of the study drug.
19. The participant has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to administration of the study drug.
20. The participant has undergone blood component collection within 2 weeks (14 days) prior to administration of the study drug.
21. The participant has any clinically significant electrocardiographic (ECG) abnormalities at the time of screening or baseline examination.
22. The participant has abnormal laboratory values that suggest a clinically significant underlying disease, or the participant has the following lab abnormalities at the time of screening or baseline examination: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 × the upper limits of normal, or differential white blood count (monocytes) < the lower limit of normal.

    The following criteria will be evaluated by laboratory tests at the screening: insulin (fasting), parathyroid hormone (PTH) (intact).
23. The participant has systolic blood pressure <80 mmHg or diastolic blood pressure <45 mmHg, or systolic blood pressure >160 mmHg or diastolic blood pressure >100 mmHg at the time of screening, baseline examination or examination prior to administration of the study drug.
24. The participant is receiving treatment for a wound and is, in the opinion of the investigator, unsuitable to participate in the study.
25. The participant is scheduled to undergo surgery within 12 weeks (84 days) after administration of the study drug.
26. In the opinion of the investigator, the participant is unlikely to comply with the protocol or is unsuitable for any other reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting One or More Treatment-emergent Adverse Events | Up to Day 37
  The adverse event is defined as any unfavorable and unintended sign, symptom, or disease that develops when a drug is administered, irrespective of the causal relationship to the drug.

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of MLN1202 | Up to Day 37
  Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Area under the serum concentration-time curve (AUC) of MLN1202 in serum | Up to Day 37
  Area under the serum concentration-time curve during a dosing interval.
Changes in serum monocyte chemoattractant protein-1 (MCP-1) concentrations | Up to Day 37
  Serum MCP-1 concentrations will be measured at each protocol-specified time point, when blood samples are collected.
Changes in monocyte count from baseline | Up to Day 37
  The absolute monocyte count will be determined at each protocol-specified time point, when blood samples are collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda
Locations (1):
- Sumida-ku, Tokyo, Japan